CLINICAL TRIAL: NCT07333404
Title: The Effects of Combined Transcranial Direct Current Stimulation and Pneumatic Compression on Selected Recovery Parameters After a 10K Run
Brief Title: Combined tDCS and Pneumatic Compression for Recovery After a 10K Run
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ramiz ARABACI, Professor, Uludag University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2025-17/11
Record Dates: First submitted 2025-12-16; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-11

CONDITIONS: Recovery Methods; Muscle Fatigue; Exercise Performance Recovery; Endurance Exercise
Keywords: master athletes; recovery; pneumatic compression; transcranial direct current stimulation; exercise performance
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Each participant will experience all four intervention conditions (transcranial direct current stimulation [tDCS], pneumatic compression [PC], combined tDCS and PC, and control) in a randomized order, with a one-week washout period between sessions to minimize carryover effects.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tDCS (Experimental): 20 minutes of transcranial direct current stimulation (tDCS) applied to the F3 and F4 regions of the brain using the Brain Premier device at 2 mA intensity.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Pneumatic Compression (PC) (Experimental): 20 minutes of sequential pneumatic compression (PC) applied to the lower limbs using the Normatec device, with compression pressure adjustable between 20 to 100 mmHg.
  Interventions: Device: Normatec Pneumatic Compression
- tDCS + PC (Experimental): Participants will receive simultaneous application of transcranial direct current stimulation (tDCS) to the F3 and F4 regions and pneumatic compression (PC) to the lower limbs for 20 minutes, combining both interventions.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Device: Normatec Pneumatic Compression
- Control (No Intervention): 20 minutes of passive rest in a semi-reclined position, no intervention applied.

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — 20 minutes of tDCS applied to F3 and F4 (left and right dorsolateral prefrontal cortex) at 2 mA using Brain Premier device in a semi-reclined position.
  Arms: tDCS; tDCS + PC
Device: Normatec Pneumatic Compression — 20 minutes of sequential pneumatic compression applied to lower limbs using Normatec device, following pressure/timing protocols (pressure 20-100 mmHg).
  Arms: Pneumatic Compression (PC); tDCS + PC

SUMMARY:
This study will examine how two recovery methods-pneumatic compression (PC) applied to the legs and transcranial direct current stimulation (tDCS) applied to the head-help athletes recover after a 10-kilometer (10K) run. It also aims to find out which methods may help master athletes recover faster, maintain performance, and reduce the risk of injury.

Men aged 40-55 who are trained long-distance runners can participate, provided they do not have medical conditions that prevent safe exercise or use of the recovery methods. Participants will run 10K and then receive one of the following interventions in a randomized order: tDCS, PC, tDCS + PC, or no intervention (control). Each participant will experience all conditions, with a one-week break between sessions. Measurements will be taken before the run, immediately after, and after the intervention, including heart rate variability, cognitive tests (Stroop Test), vertical jump, and maximal voluntary muscle contraction, during which muscle activity will be recorded using electromyography (EMG). Data will be analyzed to compare how each intervention affects recovery, including physical performance, cognitive function, and psychological state.

The study will show which methods help master runners recover faster and more effectively, provide practical strategies to improve performance and reduce injury risk, and offer information on the separate and combined effects of tDCS and PC on recovery, which could help design age-specific recovery strategies for endurance athletes.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of combined transcranial direct current stimulation (tDCS) and pneumatic compression (PC) on recovery in master male runners following a 10-kilometer run. The study also aims to examine whether these interventions can shorten recovery time and prevent performance decline after prolonged and intense exercise.

This study will be conducted as a randomized, controlled, crossover trial using a mixed experimental design. Each participant will undergo four different recovery protocols in a randomized order, with a one-week interval between sessions. Randomization will be performed using Research Randomizer, assigning participants to one of four sequences (e.g., B-A-D-C). Participants will be identified only by numerical codes to ensure blinding and maintain confidentiality. Each participant will experience all protocols, allowing within-subject comparisons and minimizing order-related bias.

The four recovery protocols are:

(A) tDCS group: transcranial direct current stimulation only (B) PC group: pneumatic compression (PC) only (C) tDCS + PC group: simultaneous application of both tDCS and PC (D) Control group: passive rest with no intervention

The tDCS and PC interventions represent the independent variables, while dependent variables include the Well-being Questionnaire (WBQ), Total Quality Recovery (TQR), heart rate variability (HRV), Stroop Test performance, vertical jump height, and maximal voluntary isometric contraction (MVIC) with electromyography (EMG) recordings.

Participants will be 35 male long-distance master runners aged 40-55 years, residing in Bursa, Turkey, with at least five years of consistent training. Participants will train five days per week for approximately 90 minutes per day and must meet aerobic fitness criteria established by the American College of Sports Medicine, including completion of an official 10-kilometer race under 50 minutes within the past six months and maintenance of a weekly running volume of 60-80 kilometers. Volunteers will be recruited from the local long-distance running community familiar to the principal investigator, Hilal Oruç Kaya.

Participants will be excluded if they have used regular medications within the last six months; consumed stimulants, caffeine, or alcohol within 24 hours prior to testing; smoke; have experienced musculoskeletal injuries within the past six months; are currently undergoing physical therapy; or have neurological conditions such as epilepsy or a history of seizures, or possess cardiac, brain, or other electronic implants. Additional exclusion criteria include open wounds or dermatological conditions on the head, circulatory disorders such as deep vein thrombosis, peripheral arterial disease, severe varicose veins, or prior exposure to tDCS or PC interventions. Participants may withdraw voluntarily, fail to attend sessions, or be removed if cardiovascular, neurological, or orthopedic complications occur during exercise or interventions, or if they experience excessive discomfort or adverse effects from the tDCS or PC procedures. Written informed consent will be obtained after participants are informed about the study's purpose, procedures, potential risks, and benefits.

Sample size was calculated using G*Power version 3.1.9.7 for repeated-measures analysis of variance with within-between interaction, assuming an effect size of f = 0.30, an alpha level of 0.05, and a statistical power of 0.80, resulting in a required sample size of 28 participants. To account for potential dropouts, a total of 35 participants will be recruited.

Screening and Familiarization Session

Participants will undergo anthropometric measurements (body mass, body fat percentage, and height) using a Tanita BC 418 MA body composition analyzer and a Seca stadiometer. Physical fitness will be evaluated using a 12-minute Cooper Test conducted on a 400-meter outdoor track under controlled environmental conditions (temperature 20-24°C, relative humidity 50-70%, wind speed ≤10 km/h). A standardized 20-minute warm-up, including jogging, accelerations, jumps, and stretching exercises, will precede the test. Distances will be recorded using a Polar V3 global positioning system (GPS) watch.

Participants will also complete a familiarization session with the 10-kilometer running course, tDCS and PC devices, the Stroop Test, MVIC procedures, and vertical jump assessments to ensure understanding of all study procedures.

Experimental Sessions

Pre-run Measurements (T1): Participants will complete the Well-being Questionnaire (WBQ) and Total Quality Recovery (TQR) scales. Heart rate (HR) and heart rate variability (HRV) will be recorded for 10 minutes using a Polar V3 GPS watch and an H10 heart rate monitor. Cognitive performance will be assessed using the Stroop Test, vertical jump height will be measured, and MVIC of the quadriceps muscles will be recorded with electromyography (EMG).

10-Kilometer Run: Participants will complete a 10-kilometer run at 75% exercise intensity calculated using the Karvonen formula. Exercise intensity will be monitored using GPS and HR data. Perceived exertion will be assessed using the Borg 20-point Rating of Perceived Exertion scale at the 5-kilometer mark and immediately after completion of the run.

Post-run Measurements (T2): All measurements obtained at T1 will be repeated immediately after the 10-kilometer run.

Interventions

Participants will be randomly assigned to one of the four recovery protocols:

tDCS: 20 minutes of 2 mA stimulation applied to the F3 and F4 regions of the dorsolateral prefrontal cortex in a semi-reclined position using the Brain Premier device

PC: 20 minutes of sequential pneumatic compression applied to the lower limbs using the Normatec pneumatic compression system, with compression pressure adjustable between 20 and 100 mmHg, following standardized pressure and timing protocols

tDCS + PC: simultaneous application of both interventions for 20 minutes

Control: passive rest in a semi-reclined position for 20 minutes

Participants in the tDCS conditions will report sensations and perceived intensity of stimulation (e.g., itching, burning, discomfort) using a structured questionnaire.

Post-intervention Measurements (T3): All measurements obtained at T1 will be repeated immediately after the intervention.

Outcome Measures

Subjective recovery measures: Well-being Questionnaire (WBQ) and Total Quality Recovery (TQR)

Autonomic measures: heart rate variability (HRV) and GPS-derived data

Cognitive performance assessed using the Stroop Test

Vertical jump height assessed using the My Jump application

MVIC of the quadriceps muscles recorded with electromyography (EMG) following the Surface Electromyography for the Non-Invasive Assessment of Muscles (SENIAM) guidelines

Statistical Analysis

Data will be analyzed using IBM SPSS Statistics version 29. Normality will be assessed using the Shapiro-Wilk test, homogeneity of variances using Levene's test, and sphericity using Mauchly's test. A two-way repeated-measures analysis of variance (4 Time × 4 Condition) will be used to evaluate interaction effects, with Bonferroni-adjusted post hoc comparisons applied when appropriate. Effect sizes will be reported using partial eta squared (ηp²), with values of >0.01 considered small, >0.06 medium, and >0.14 large. Statistical significance will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria

* Age 40 to 55 years
* Completion of an official 10-kilometer race in under 50 minutes within the last six months
* Regular training 5 days per week, 90 minutes per day
* Weekly running volume of 60-80 kilometers
* Aerobic fitness ≥ 80% according to American College of Sports Medicine (ACSM) guidelines

Exclusion Criteria

* Use of regular medications within the last six months
* Consumption of stimulants, caffeine, or alcohol within 24 hours prior to testing
* Smoking
* Musculoskeletal injuries within the last six months
* Participation in current physical therapy programs
* Epilepsy or history of seizures
* Cardiac, brain, or other electronic implants
* Open wounds or dermatological conditions on the head
* Circulatory disorders, including deep vein thrombosis, peripheral arterial disease, or severe varicose veins
* Previous exposure to transcranial direct current stimulation (tDCS) or pneumatic compression (PC) interventions

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-05-27 (Estimated); Study Completion 2026-06-27 (Estimated)

PRIMARY OUTCOMES:
Maximal Voluntary Isometric Contraction (MVIC) | Assessments will be performed immediately before the 10-kilometer run, immediately after completion of the 10-kilometer run, and immediately after the recovery intervention.
  Maximal voluntary isometric contraction (MVIC) of the quadriceps muscles (vastus lateralis, rectus femoris, and vastus medialis) will be measured using surface electromyography (EMG) to assess neuromuscular function and fatigue. Participants will perform three contractions lasting 3 to 5 seconds each, with 60-second rest intervals, while seated with the knee and hip joints positioned at 90 degrees.
Heart Rate Variability (HRV) | Immediately before 10K run, immediately after 10K run, immediately after recovery intervention
  Heart rate variability will be measured using the Polar Vantage V3 GPS watch with H10 heart rate sensor to assess autonomic nervous system responses to exercise and recovery interventions. HRV parameters will be analyzed to evaluate physiological stress and recovery. Measurements will be recorded at rest for 5 minutes in a seated position.
Cognitive Performance: Stroop Test | Immediately before 10K run, immediately after 10K run, immediately after recovery intervention
  Cognitive performance will be assessed using the computerized Stroop Test. Participants will respond to color-word stimuli where the color of the word may be congruent or incongruent with the written word. Reaction time and accuracy will be recorded to evaluate cognitive function and executive control in response to exercise and recovery interventions.

SECONDARY OUTCOMES:
Total Quality Recovery (TQR) | Immediately before the 10-kilometer run (T1), immediately after the 10-kilometer run (T2), and immediately after the recovery intervention (T3).
  Participants will self-report perceived recovery using the Total Quality of Recovery scale, assessing overall recovery status after exercise and recovery interventions. Scores range from 1 to 10, with higher scores indicating better recovery quality.
Well-Being Questionnaire (WBQ) | Immediately before the 10-kilometer run (T1), immediately after the 10-kilometer run (T2), and immediately after the recovery intervention (T3).
  Participants will complete the Well-Being Questionnaire to evaluate subjective measures of mood, fatigue, and general well-being in response to exercise and recovery interventions. Scores range from 1 to 5, with higher scores indicating better well-being.
Vertical Jump | Immediately before 10K run, immediately after 10K run, immediately after recovery intervention
  Participants will perform three maximum effort vertical jumps at one-minute intervals. Jump height will be measured using the MyJump app to assess neuromuscular performance after exercise and recovery interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University, Faculty of Sport Sciences, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared due to privacy concerns and the study's data management plan. All data will be used solely for the purposes of the current research and will not be made available to external researchers.

REFERENCES:
- [Result] Goncalves DS, Moscaleski LA, da Silva GM, Morgans R, Okano AH, Moreira A. The Effect of Combined Transcranial Direct Current Stimulation and Pneumatic Compression as Part of a Comprehensive Recovery Strategy in Professional Male Top-Level Soccer Players. J Strength Cond Res. 2024 Sep 1;38(9):1658-1666. doi: 10.1519/JSC.0000000000004844. Epub 2024 Jul 23. PMID 39074250
- [Result] Shiravand F, Motamedi P, Amani-Shalamzari S, Amiri E, da Silva Machado DG. Effect of repeated sessions of transcranial direct current stimulation on subjective and objective measures of recovery and performance in soccer players following a soccer match simulation. Sci Rep. 2024 Sep 6;14(1):20809. doi: 10.1038/s41598-024-71701-y. PMID 39242725

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT07333404/Prot_SAP_000.pdf
  • Informed Consent Form (2025-12-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT07333404/ICF_001.pdf